CLINICAL TRIAL: NCT03678935
Title: Effect of Fermentable Oligo-, di-, and Monosaccharides and Polyols (FODMAP) Restriction on Persistent GI-symptoms in Coeliac Patients
Brief Title: Effect of FODMAP Restriction on Persistent GI-symptoms in Coeliac Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Responsible Party: Principal Investigator, Knut E. A. Lundin, Professor medicine, Oslo University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2018/1055
Record Dates: First submitted 2018-09-17; First posted 2018-09-20 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: Celiac Disease; Irritable Bowel Syndrome; Diet Modification; Gluten Sensitivity
Keywords: Celiac disease; Irritable bowel syndrome
MeSH Terms: conditions — Celiac Disease; Irritable Bowel Syndrome | interventions — FODMAP Diet

STUDY DESIGN:
Intervention Model Description: The intervention group receives advice on following the low-FODMAP diet, and the control group follows their regular gluten free diet.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low FODMAP diet (LFD) (Active Comparator): The LFD wil receive advice on how to follow a low FODMAP diet. They wil follow this diet for 4 weeks. Thereafter they receive advice on how to reintroduce high FODMAPs again.
  Interventions: Other: Low FODMAP diet
- Control (No Intervention): Control group. Participants follow their regular gluten-free diet (GFD), with no changes to their diet. They wil receive the same dietary advice as the LFD-group after the 4-week study.

INTERVENTIONS:
Other: Low FODMAP diet — The intervention group follows the low FODMAP diet for 4 weeks.
  Arms: Low FODMAP diet (LFD)

SUMMARY:
The first aim of the study is to investigate the prevalence of persistent gastrointestinal symptoms and compliance with gluten-free diet and the intake of FODMAP in adult celiac patients.

A web-based survey wil be performed and thereafter a randomized controlled trial to test the effect of a FODMAP reduction in patients with celiac disease with irritable bowel-like symptoms.

DETAILED DESCRIPTION:
Effect of FODMAP reduction in patients with celiac disease. Celiac disease is an immune-mediated disease that causes damage to the intestines. The condition affects 1-2% of the population, and the incidence is increasing. Treatment with gluten-free diet usually produces good results, yet there are many patients who have persistent gastrointestinal symptoms. Studies indicate that this applies to as many as 20%, but the situation in Norway in unknown. Nor is it known why somebody has persistent gastro- intestinal complaints. It may be due to difficulty following the diet or what is called irritable bowel syndrome (IBS), which is a fairly common condition in the population.

It has been shown that people with IBS can benefit from a diet with reduced FODMAP content. The term FODMAP is an acronym for: Fermentable Oligo, Di-, Monosaccharides and Polyols. It is a type of carbohydrate that is not absorbed in the large intestine, but continues to the colon where they are fermented by the bacteria. Example of foods with a high content of FODMAP is wheat, onion, garlic, parsley, apples, pears, mango, beans, honey and milk. It is not known whether celiac patients with persistent symptoms will have the beneficial effect of low FODMAP diet.

In this study, investigators want to study the prevalence of persistent gastrointestinal symptoms and compliance with gluten-free diet and the intake of FODMAP in adult celiac patients. Members of the Norwegian coeliac organization will be invited to participate in the study. A web-based questionnaire is used to make it easy for members to respond.

Participants who report persistent gastrointestinal intestinal symptoms will then be invited to a randomized and controlled study. They will be divided into two groups where one group will be advised to reduce the intake of FODMAP and the other group will be advised to follow a strict gluten-free diet. Participants will record stomach and intestinal complaints before and after four weeks with study sites. Investigators will find out whether there is a difference between gastric and intestinal complaints between the two groups. Blood- and feces samples will also be collected.

The results will provide new knowledge about how to adapt dietary advice to celiac patients with persistent gastrointestinal complaints, and hopefully help them to a better quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Coeliac disease
* Adherent to GFD for at least 12 months
* Strictly adherent to GFD
* Normal coeliac disease (CD) serology and duodenal biopsy (Marsh 0-1)
* Persistent GI-symptoms defined by GSRS-IBS score of 30 or more
* Living less than 2 hour from study centre

Exclusion Criteria:

* Pregnancy or lactating women
* Use of immunomodulating drugs in the last 3 months
* Use of anti-inflammatory drugs in the last 3 months
* Use of antacid drugs in the last 2 months
* Ongoing infection (mild infection such as upper airway infection is ok)
* Other chronical bowel disorder (except for IBS)
* Previous tried the LFD with guidance of a dietician

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2025-07-28 (Actual); Study Completion 2025-07-28 (Actual)

PRIMARY OUTCOMES:
Change in gastrointestinal symptoms | 4 weeks
  Measured by score in gastrointestinal symptom rating scale for irritable bowel syndrome (GSRS-IBS). The scoring is based on a 7-grade Likert scale in which 1 point indicates no symptoms and 7 points the most severe gastrointestinal symptoms. The total score in the gastrointestinal symptom rating scale for irritable bowel syndrome is calculated as a mean value of all 13 items. The maximum score is 91 and the minimum score is 13. A higher score means more severe symptoms. A score higher than 1 standard deviation (SD, 0.66 points) compared to the control mean are considered to have increased gastrointestinal symptoms.

SECONDARY OUTCOMES:
Changes in biomarkers like faecal microbiota | 4 weeks
  Altered faecal microbiota diversity, measured as a change in diversity and/or abundance or strains from baseline and after 4 weeks on a low FODMAP diet.
Quality of Life in patients with coeliac disease: Short form- 36 (SF-36) | 4 weeks
  Changes in short form-36 (SF-36) as a measure of quality of life. SF-36 covers four physical health perceptions (physical functioning, role limitations because of physical health problems, bodily pain, and general health) and four mental health concepts (vitality, social functioning, role limitations because of personal or emotional problems, and mental health perceptions). Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The range of score is 0 to 100, where a higher score means better quality of life and the lower the score the more disability. A total score for mental health and physical health is calculated as an average of the subscales, with a range from 0 to 100. Here also the higher the score the better quality of life. The standardized combined scores in several populations have a mean of 50 and standard deviation 10. The scoring wil be performed as in the SF-36 scoring manual.

CONTACTS AND LOCATIONS:
Overall Officials: Knut Lundin, Professor, Principal Investigator — Oslo University hospital and University of Oslo
Locations (1):
- Rikshospitalet-Radiumhospitalet HF, Oslo University Hospital, Oslo, Postboks PB 4950 Nydalen, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Herfindal AM, van Megen F, Gilde MKO, Valeur J, Rudi K, Skodje GI, Lundin KEA, Henriksen C, Bohn SK. Effects of a low FODMAP diet on gut microbiota in individuals with treated coeliac disease having persistent gastrointestinal symptoms - a randomised controlled trial. Br J Nutr. 2023 Dec 28;130(12):2061-2075. doi: 10.1017/S0007114523001253. Epub 2023 Jun 5. PMID 37272479
- [Result] van Megen F, Skodje GI, Lergenmuller S, Zuhlke S, Aabakken L, Veierod MB, Henriksen C, Lundin KEA. A Low FODMAP Diet Reduces Symptoms in Treated Celiac Patients With Ongoing Symptoms-A Randomized Controlled Trial. Clin Gastroenterol Hepatol. 2022 Oct;20(10):2258-2266.e3. doi: 10.1016/j.cgh.2022.01.011. Epub 2022 Jan 17. PMID 35051648
- [Result] van Megen F, Fossli M, Skodje GI, Carlsen MH, Andersen LF, Veierod MB, Lundin KEA, Henriksen C. Nutritional assessment of women with celiac disease compared to the general population. Clin Nutr ESPEN. 2023 Apr;54:251-257. doi: 10.1016/j.clnesp.2023.01.031. Epub 2023 Feb 2. PMID 36963870
- [Result] Skodje GI, van Megen F, Stendahl M, Henriksen C, Lundin KEA, Veierod MB. Detection of gluten immunogenic peptides and the Celiac Disease Adherence Test to monitor gluten-free diet: a pilot study. Eur J Clin Nutr. 2022 Jun;76(6):902-903. doi: 10.1038/s41430-021-01054-6. Epub 2022 Jan 10. PMID 35001079
- [Result] van Megen F, Skodje GI, Stendahl M, Veierod MB, Lundin KEA, Henriksen C. High disease burden in treated celiac patients - a web-based survey. Scand J Gastroenterol. 2021 Aug;56(8):882-888. doi: 10.1080/00365521.2021.1930146. Epub 2021 May 30. PMID 34057009

DOCUMENTS (1):
  • Study Protocol (2018-06-01): https://cdn.clinicaltrials.gov/large-docs/35/NCT03678935/Prot_002.pdf